CLINICAL TRIAL: NCT04763759
Title: A Phase 1, Blinded, Single Ascending Dose Study to Evaluate Safety, Pharmacokinetics, and Activity of TRL1068 in Subjects with Prosthetic Joint Infection of the Knee or Hip, Undergoing Primary Two Stage Exchange Arthroplasty
Brief Title: Study to Evaluate Safety and Activity of TRL1068 in Prosthetic Joint Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trellis Bioscience LLC (Industry)
Collaborators: University of California, Los Angeles (Other); Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); Sinai Hospital of Baltimore (Other); Gulfcoast Research Institute (Unknown); Phoenix Clinical Research (Other); University of Florida (Other); University of Alabama at Birmingham (Other); The Methodist Hospital Research Institute (Other); University of Virginia (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRL1068-101
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Prosthetic Joint Infection
Keywords: biofilm; antibiotic-resistant infections
MeSH Terms: interventions — TRL1068

STUDY DESIGN:
Intervention Model Description: Phase 1, Double-Blinded, Single Ascending Dose Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind and placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1- 6mg/kg (Experimental): Randomized 3:1 (TRL1068:placebo) via IV infusion
  Interventions: Drug: TRL1068, a human monoclonal antibody
- Dose Level 2- 15mg/kg (Experimental): Randomized 5:2 (TRL1068:placebo) via IV infusion
  Interventions: Drug: TRL1068, a human monoclonal antibody
- Dose Level 3- 30 mg/kg (Experimental): Randomized 5:2 (TRL1068:placebo) via IV infusion
  Interventions: Drug: TRL1068, a human monoclonal antibody

INTERVENTIONS:
Drug: TRL1068, a human monoclonal antibody — A human IgG1κ (G1m1,17 (z,a); Km3 allotype) monoclonal antibody

SUMMARY:
TRL1068 is expected to eliminate the pathogen-protecting biofilm in the prosthetic joint and surrounding tissue, thus making these pathogens substantially more susceptible to established antibiotic treatment regimens. This initial study is designed to assess overall safety and pharmacokinetics (PK) of TRL1068. The overall goal of the development program is to demonstrate that TRL1068 can facilitate effectiveness of a single stage joint replacement or preservation of the original infected prosthetic joint in a substantial proportion of patients with PJI.

DETAILED DESCRIPTION:
Approximately 75% of all clinically significant human infections are estimated to be biofilm-related. Prosthetic joint infections are a classical example of difficult to eradicate infections associated with biofilm. Most Prosthetic Joint Infection (PJI) cases are caused by staphylococcal species (~70%) with an increasing number being antibiotic-resistant (MRSA). In the US, two-stage revision is the standard of care for replacement of an infected prosthetic joint, and is associated with substantial costs and prolonged immobility. TRL1068 is a fully human antibody that has been shown in pre-clinical studies to disrupt biofilm. TRL1068 targets a highly conserved epitope on the DNABII family of bacterial DNA binding proteins that includes histone-like (HU) and integration host factor (IHF) proteins of clinically relevant Gram-positive and Gram-negative bacteria. The DNABII epitope bound by TRL1068 has no homologs in the human proteome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PJI of the knee or hip
* Identified pathogen(s) must be susceptible to antibiotic regimen
* Planned/scheduled for primary two-stage exchange arthroplasty
* BMI < 40 kg/m²
* Willing and able to provide written informed consent
* Willing to perform and comply with all study procedures including attending clinic visits as scheduled.
* Men and women of child bearing potential (WOCBP) must be willing to practice a highly effective method of contraception

Exclusion Criteria:

* Evidence of active infection other than bacterial PJI of the knee or hip
* Inability to receive or intolerant to pathogen-appropriate systemic or oral antibiotic therapy
* Chronic obstructive pulmonary disease (COPD)
* Child-Pugh score > 6
* Congestive heart failure
* Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids
* Active malignancy, or history of malignancy or chemotherapy within the past 2 years
* Active or history of autoimmune disease
* Uncontrolled diabetes, defined as hemoglobin A1c > 7.4%
* Clinically significant abnormality on electrocardiogram (ECG) that would preclude subject from undergoing two-stage exchange arthroplasty
* Clinically significant serum chemistry or hematology abnormalities
* Any acute illness within 14 days of Day 1 that could confound the evaluation of safety evaluation
* Known or suspected intolerance or hypersensitivity to any biologic medication
* Received a therapeutic antibody or biologic within the 6 months prior to Screening
* Positive serum test for pregnancy, pregnant, or nursing women
* Positive reverse transcription polymerase chain reaction (RT -PCR) or alternative (antigen) test for acute respiratory syndrome coronavirus 2
* History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the subject's ability to comply with the study requirements
* Any other comorbidity or condition that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Abnormal Physical Examination Findings | 16 weeks
  clinically significant abnormal physical exam findings will be reviewed
Incidence of Abnormal Serum Chemistries and Hematology | 16 weeks
  clinically significant abnormal laboratory results will be reviewed
Incidence of Abnormal Vital Signs (Temperature) | 16 weeks
  clinically significant abnormal temperatures will be reviewed
Incidence of Abnormal Vital Signs (Blood Pressure) | 16 weeks
  clinically significant abnormal blood pressures will be reviewed
Incidence of Abnormal Vital Signs (Heart Rate) | 16 weeks
  clinically significant abnormal heart rates will be reviewed
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 24 weeks
  mortality and any other reported AEs and SAEs will be reviewed

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) of a single IV infusion of TRL1068 | 16 weeks
  Serum and synovial concentrations of TRL1068 will be determined by ELISA
Measure TRL1068 levels in synovial fluid on Day 8 and compare with plasma PK | 1 week
  Serum and synovial concentrations of TRL1068 will be determined by ELISA
Assess the pharmacodynamics (PD) of TRL1068 (Colony Forming Units (CFUs) prosthesis) | 1 week
  Number of CFUs from sonicated prosthetic device
Assess the pharmacodynamics (PD) of TRL1068 (CFUs spacer) | 12 weeks
  Number of CFUs from sonicated orthopedic spacer
Assess the pharmacodynamics (PD) of TRL1068 (CRP) | 16 weeks
  Inflammatory biomarker CRP
Assess the pharmacodynamics (PD) of TRL1068 (ESR) | 16 weeks
  Inflammatory biomarker ESR
Assess the pharmacodynamics (PD) of TRL1068 (IL-6) | 16 weeks
  Inflammatory biomarker IL-6
Assess the pharmacodynamics (PD) of TRL1068 (IL-10) | 16 weeks
  Inflammatory biomarker IL-10
Assess the pharmacodynamics (PD) of TRL1068 (reinfection) | 24 weeks
  Assessment for reinfection including need for further surgical interventions and overall outcome
Assess the immunogenicity of TRL1068 as measured by anti-drug antibodies (ADAs) | 16 weeks
  Anti-drug antibodies (ADA), i.e. anti-TRL1068 antibodies in serum will determined by electrochemiluminescence assay.

OTHER OUTCOMES:
Exploratory outcome measure to determine CFUs | 12 weeks
  The number of subjects with Colony Forming Units (CFUs) per mL ≥ 1 from sonicated prosthetic devices from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to determine inflammation (CRP) | 16 weeks
  The mean levels of C reactive protein (CRP) from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to determine inflammation (ESR) | 16 weeks
  The mean levels of erythrocyte sedimentation rate (ESR) from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to determine inflammation (IL-6) | 16 weeks
  The mean levels of Interleukin-6 (IL-6) from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to determine inflammation (IL-10) | 16 weeks
  The mean levels of Interleukin-10 (IL-10) from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to determine infection in synovial fluid | 1 week
  The number of subjects with CFUs/mL ≥ 1 from the synovial fluid from placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure inflammation in the synovial fluid | 1 week
  The mean synovial fluid total leukocyte cell counts of the consolidated placebo and TRL1068 treated groups will be compared.
Exploratory outcome measure to assess quality of life | 24 weeks
  Patient-Reported Outcomes Measurement Information System - Physical Function (PROMIS-PF) Short Form 6b from placebo and TRL1068 treated groups will be compared. This questionnaire has a score range from 6-30, with higher scores indicating higher functioning than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bernthal, MD, Principal Investigator — University of California, Los Angeles; Janet Conway, MD, Principal Investigator — Sinai Hospital of Baltimore; Edward Stolarski, MD, Principal Investigator — Gulfcoast Research Institute; Richard Berkowitz, MD, Principal Investigator — Phoenix Clinical Research; Luis Pulido, MD, Principal Investigator — University of Florida; Sameer Naranje, MD, Principal Investigator — University of Alabama at Birmingham; Stephen Incavo, MD, Principal Investigator — The Methodist Hospital Research Institute; Ian Duensing, MD, Principal Investigator — UVA; Daniel Oakes, MD, Principal Investigator — University of Southern California
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - USC, Los Angeles, California
  - UCLA, Santa Monica, California
  - University of Florida, Gainesville, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Houston Methodist Research Institute, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
The study results have been published.

REFERENCES:
- [Background] Conway J, Delanois RE, Mont MA, Stavrakis A, McPherson E, Stolarski E, Incavo S, Oakes D, Salvagno R, Adams JS, Kisch-Hancock A, Tenorio E, Leighton A, Ryser S, Kauvar LM, Bernthal NM. Phase 1 study of the pharmacokinetics and clinical proof-of-concept activity of a biofilm-disrupting human monoclonal antibody in patients with chronic prosthetic joint infection of the knee or hip. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0065524. doi: 10.1128/aac.00655-24. Epub 2024 Jul 16. PMID 39012102
- [Background] Estelles A, Woischnig AK, Liu K, Stephenson R, Lomongsod E, Nguyen D, Zhang J, Heidecker M, Yang Y, Simon RJ, Tenorio E, Ellsworth S, Leighton A, Ryser S, Gremmelmaier NK, Kauvar LM. A High-Affinity Native Human Antibody Disrupts Biofilm from Staphylococcus aureus Bacteria and Potentiates Antibiotic Efficacy in a Mouse Implant Infection Model. Antimicrob Agents Chemother. 2016 Mar 25;60(4):2292-301. doi: 10.1128/AAC.02588-15. Print 2016 Apr. PMID 26833157
- [Background] Xiong YQ, Estelles A, Li L, Abdelhady W, Gonzales R, Bayer AS, Tenorio E, Leighton A, Ryser S, Kauvar LM. A Human Biofilm-Disrupting Monoclonal Antibody Potentiates Antibiotic Efficacy in Rodent Models of both Staphylococcus aureus and Acinetobacter baumannii Infections. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00904-17. doi: 10.1128/AAC.00904-17. Print 2017 Oct. PMID 28717038